CLINICAL TRIAL: NCT03269968
Title: Use of Negative Pressure Wound Therapy in Morbidly Obese Women After Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Amenity Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-137
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-06

CONDITIONS: Obesity, Morbid; Wound Infection; Wound Complication
MeSH Terms: conditions — Obesity, Morbid; Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Study participants will be enrolled in a 1:1 ratio to either Negative Pressure Wound Therapy or standard dressing. Randomization will occur prior to delivery using a computer randomization system.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative pressure wound therapy (NPWT) (Experimental): Women receiving NPWT will have a PREVENA Incision Management Therapy System applied directly onto their skin over the closed incision after delivery.
  Interventions: Device: Negative pressure wound therapy (PREVENA Incision Management Therapy System)
- Standard dressing (Placebo Comparator): Standard dressing
  Interventions: Device: Standard dressing

INTERVENTIONS:
Device: Negative pressure wound therapy (PREVENA Incision Management Therapy System) — After cesarean delivery, women in the intervention group will receive PREVENA Incision Management Therapy System.
  Arms: Negative pressure wound therapy (NPWT)
Device: Standard dressing — After cesarean delivery, women in the intervention group will receive standard dressing.
  Arms: Standard dressing

SUMMARY:
Obese women are more likely have a cesarean delivery and develop subsequent wound complications than normal weight women. Negative pressure wound therapy (NPWT) has been shown to improve surgical wound healing, but this device has not been adequately studied in cesarean deliveries. The aim of our study is to determine the efficacy of NPWT in morbidly obese women after cesarean delivery.

Investigators will be randomizing women with a BMI > 40 kg/m2 in a 1:1 ratio to either NPWT (the PREVENA Incision management therapy system Pre 1001 Us) or standard dressing after their cesarean delivery at MedStar Washington Hospital Center. The NPWT will be left in place for a minimum of four days but not to exceed seven days. The standard dressing is typically removed on postoperative day one or two. The primary outcome is a wound complication defined as the formation of a wound infection, seroma, hematoma, separation, or dehiscence from delivery to 4 weeks postpartum. Investigators will also administer a patient satisfaction survey regarding their wound healing experience.

DETAILED DESCRIPTION:
Obese women are more likely to be delivered by cesarean than normal weight women and are at increased risk for operative morbidity including wound complications. Negative pressure wound therapy (NPWT) has been shown to improve wound healing, decrease the rate of surgical site infection, sero-hematoma formation, and reoperation rates. The potential benefit of NPWT in high-risk wounds after cesarean delivery is unclear. Investigators propose conducting a single-site randomized controlled trial to examine the efficacy of NPWT after cesarean delivery in morbidly obese women (BMI ≥ 40 kg/m2).

Specific aims of the study include determining if NPWT used in morbidly obese women after cesarean delivery improves postoperative wound complication rate and to assess patient satisfaction with NPWT. The primary outcome is a composite wound complication rate defined as having one of the following occur within four weeks of delivery: wound infection, seroma, hematoma, separation, or dehiscence.

Participants will be randomized in a 1:1 ratio to either NPWT or standard surgical dressing. Women receiving NWPT will have a PREVENA Incision Management Therapy System applied directly onto their skin over the closed incision after delivery. Women randomized to the standard surgical dressing will have a TELFA non-adhesive dressing with a 3M Tegaderm transparent film adhesive dressing. In addition, an abdominal pad (ABD) with foam tape may be applied to provide additional pressure if needed.

The wound will be assessed at the time of dressing removal or hospital discharge and at four weeks postoperative. Participants will also take a patient satisfaction survey regarding wound healing experience at four-week follow-up. For the study, investigators are planning to enroll 482 patients (241 per arm) to demonstrate a decrease in the wound complication rate by 50%. This study will help clinicians better manage obese women in pregnancy and hopefully improve wound outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≥40 kg/m2 at time of delivery
* Delivered by cesarean delivery
* 18 years or later

Exclusion Criteria:

* Chorioamnionitis
* Silver allergy
* Inability to follow up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 25 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachael T Overcash, MD, MPH, Principal Investigator — Medstar Health Research Institute; Iqbal N Iqbal, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated due to insufficient enrollment. No study data are available.
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy (NPWT) | Standard Dressing
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated due to insufficient enrollment. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Therapy (NPWT) | Standard Dressing | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]
Parity

OUTCOME MEASURES:

1. Primary Outcome: Composite Wound Complication
Description: Any of wound infection, seroma/hematoma, wound separation >1 cm, and wound dehiscence
Time Frame: Four weeks postpartum
Population: The study was terminated due to insufficient enrollment. No study data are available.
Arm/Group | Negative Pressure Wound Therapy (NPWT) | Standard Dressing
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Survey
Description: Through patient surveys administered prior to hospital discharge and at four weeks post-operative investigators will evaluate patient satisfaction with wound healing. Satisfactory measures will include how well participants think incision healed mobility after surgery, pain control, and the incision's appearance. Patients were also asked if they had emergency room visits or hospital readmissions. For patients who received NPWT investigators will assess the ease of use, comfort, and perception of its efficacy.
Time Frame: Four weeks postpartum
Population: The study was terminated due to insufficient enrollment. No study data are available.
Arm/Group | Negative Pressure Wound Therapy (NPWT) | Standard Dressing
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Demographic Data
Description: Age, race/ethnicity, parity
Time Frame: At time time of admission
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Maternal Body Mass Index
Description: Prepregnancy and at the time of delivery
Time Frame: At time time of admission
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Gestational Age at Delivery
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At time time of admission
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Maternal Comorbidities
Description: Renal disease, hypertension, diabetes, psychiatric history, sleep apnea, history of venous thromboembolism
Time Frame: At time time of admission
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Antenatal Complications
Description: Gestational diabetes, preeclampsia
Time Frame: At time time of admission
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Number of Previous Cesarean Deliveries
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At time time of admission
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Indication for Cesarean Delivery
Description: Failed induction, arrest of active phase, arrest of descent, malpresentation, repeat cesarean delivery, desired cesarean
Time Frame: At time time of cesarean delivery
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Reason for Admission
Description: Spontaneous labor, rupture of membranes, induction of labor, scheduled cesarean delivery, fetal condition (oligohydroamnios, growth restriction, non reassuring fetal heart tracing)
Time Frame: At the time of admission
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Labor Duration
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Endometritis
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: Four weeks postpartum
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Length of Rupture of Membranes
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Operative Time
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Intraoperative Complication
Description: Postpartum hemorrhage, transfusion, ureteral injury, bladder injury, B-lynch suture, and hysterectomy
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Type of Skin Incision
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Type of Uterine Incision
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Type of Fascia Closure
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Type of Subcutaneous Closure
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Administration of Preoperative Antibiotics
Description: Cefazolin, Azithromycin, Clindamycin, Gentamicin, and other
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Quantitative Blood Loss
Description: We were unable to adequately recruit for this study. Study was closed.
Time Frame: At the time of cesarean delivery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The study was terminated due to insufficient enrollment. No study data are available.
Description: The study was terminated due to insufficient enrollment. No study data are available.
Arm/Group | Negative Pressure Wound Therapy (NPWT) | Standard Dressing
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03269968/Prot_ICF_000.pdf